CLINICAL TRIAL: NCT04584723
Title: Outcomes of Microsurgical Reconstruction in the Elderly Patient in a Private Practice Setting in México City: Case Series
Brief Title: Microsurgery in the Elderly in a Private Practice Setting
Status: Completed | Type: Observational
Sponsor: Hospital Angeles del Pedregal (Other)
Responsible Party: Principal Investigator, javier lopez, Principal investigator, Plastic and reconstructive surgeon staff, MBA, FACS, Hospital Angeles del Pedregal
Other Study IDs: Elderly
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Aged; Microsurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation of flap survival and complications — We will report the flap survival and complications in this population group underwent to microsurgical procedures in a private practice setting

SUMMARY:
This study reports the experience in free tissue transfer in the elderly population by a single surgeon in the private practice setting in Mexico city and the potential criticism that could arise from adverse events in lower-volume practice situations will be addressed. Investigator will answer the question about the age as the variable of interest in this series in which age was not a factor in deciding reconstructive methods, and examine complication rates.

DETAILED DESCRIPTION:
Investigators will evaluate the outcomes of 17 flaps in 14 patients who required microsurgical reconstruction with free flaps and microvascular vessels anastomosis. All patients more than 65 years old. Demographic data will be reported as: obesity, American Society of Anesthesiology (asa) level, radiotherapy, combined surgery. And the results of investigation will include: Flap survival, local complications, systemic complications, re-interventions, 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Elderly population, defined as more than 65 years old
* Patients underwent to free flap microsurgical procedures.
* Complete files
* Patient acceptance to participate

Exclusion Criteria:

* Lost follow up

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients more than 65 years old, with indications for a free flap reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Flap survival | 1 month
  Evaluation of success of microsurgical free flap. Flap necrosis or not
Complications | 1 month
  Report the number and type of local and systemic complications in this microsurgical procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Angeles Pedregal, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
We will share, age, American society of anesthesiology (ASA) level, Obesity, radiotherapy associated. And the results of flap survival, type of complications including local and systemic.